CLINICAL TRIAL: NCT07253233
Title: A Prospective, Single-center, Single-arm Clinical Study Protocol on the Treatment of Spinal Cord Injury Using Autologous Concentrated Growth Factors
Brief Title: Treatment of Spinal Cord Injury Using Autologous Concentrated Growth Factors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Limin Rong, President, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACGF-SCI
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; growth factors; autologous
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the treatment of spinal cord injury using autologous concentrated growth factors (Experimental)
  Interventions: Biological: Concentrated Growth Factors (CGF)

INTERVENTIONS:
Biological: Concentrated Growth Factors (CGF) — Concentrated Growth Factors (CGF) have garnered significant attention owing to their distinct biological properties . CGF is a concentrated autologous platelet-rich fibrin matrix derived from centrifuged venous blood, containing high levels of bioactive growth factors, including platelet-derived growth factor (PDGF), transforming growth factor-β (TGF-β), vascular endothelial growth factor (VEGF), and insulin-like growth factor (IGF). These growth factors play pivotal roles in promoting angiogenesis, modulating inflammatory responses, and stimulating cellular proliferation and differentiation. Evidence suggests that CGF not only enhances the local microenvironment at the site of injury but also promotes neural repair by activating endogenous neural stem cells and supporting axonal regeneration, thereby offering a promising multi-target therapeutic approach for spinal cord injury recovery.

SUMMARY:
Spinal cord injury (SCI) is a severe disorder of the central nervous system, and effective clinical management remains a significant global challenge. Current therapeutic approaches can only partially restore neurological function, leaving the majority of individuals with SCI facing profound and lifelong disabilities. The Department of Spine Surgery at the Third Affiliated Hospital of Sun Yat-sen University is conducting a clinical study on the use of autologous concentrated growth factors for the treatment of spinal cord injury, with the aim of developing a novel and effective clinical intervention strategy.

DETAILED DESCRIPTION:
Research Objective: To evaluate the clinical efficacy of autologous concentrated growth factors (Concentrated Growth Factors, CGF) in promoting the recovery of motor, sensory, and autonomic functions in individuals with spinal cord injury (SCI), and to investigate the underlying mechanisms through which CGF contributes to functional restoration of the injured spinal cord.

Study Design: A prospective, single-center, single-arm clinical trial. Study Population: Individuals diagnosed with spinal cord injury who meet predefined inclusion criteria.

Intervention: Eligible participants will receive autologous concentrated growth factor biofilm implantation at the site of spinal cord injury, in conjunction with standard rehabilitation therapy. Participants will undergo structured follow-up assessments at 1, 3, and 6 months post-intervention; an additional follow-up at 12 months will be conducted as a long-term observational time point.

Outcome Measures:

Primary Outcome Measure: Change in ASIA motor score from baseline to each follow-up visit.

Secondary Outcome Measures: ASIA sensory scores, International Association for Neurorestoration-Spinal Cord Injury Functional Rating Scale (IANR-SCIFRS), Spinal Cord Independence Measure-III (SCIM III), 10-meter Walk Test (10MWT), International Standards for Autonomic Function after SCI (ISAFSCI), Hospital Anxiety and Depression Scale (HADS), bladder function assessment (Geffner scale), bowel function assessment (Neurogenic Bowel Dysfunction Score, NBD), muscle tone evaluation (Modified Ashworth Scale), spasticity assessment (Penn Spasm Frequency Scale), somatosensory evoked potentials (SEP), and multimodal magnetic resonance imaging (MRI) of the brain and spinal cord.

Sample Size: This is an exploratory pilot study designed to enroll 10 participants.

Statistical Analysis Plan: The full analysis set (FAS), per-protocol set (PPS), and safety analysis set will be established. Descriptive statistics will include data distribution assessment (normality testing), summary of baseline characteristics, handling of missing data, and dropout analysis. Inferential statistical analyses will include within-group comparisons over time using appropriate longitudinal models, assessment of potential center effects (if applicable), safety profile evaluation, and exploratory logistic regression analyses to identify potential predictors of response.

ELIGIBILITY:
Inclusion Criteria:

* Chinese citizens, aged 18-60;

  * Spinal cord injury caused by trauma;

    * ASIA spinal cord injury grade C-D; ④ Duration of the disease: Acute, subacute and chronic spinal cord injuries are all acceptable; ⑤ Cooperate to complete the follow-up.

Exclusion Criteria:

* Severe systemic diseases;

  * Joint contractures;

    * Having hematological diseases, autoimmune diseases and infectious diseases;

      * Prohibited conditions for magnetic resonance imaging and electrophysiological examinations（For example：intracranial metal implants， cardiac stents, spinal stimulators, spinal internal fixators)；

        * Severe anxiety/depression/manic states， or diagnosed with mental illness or epilepsy； ⑥ Spinal cord injury caused by myelitis， multiple sclerosis， or spinal tumors；

          * Complicated with bleeding disorders or coagulation dysfunction；

            * Individuals with osteoporosis and a high risk of pathological fractures； ⑨ Poor compliance， or unable to correctly understand and cooperate to complete follow-up； ⑩ Pregnant or lactating women； ⑪ Those who have received other spinal cord injury intervention treatments such as stem cells or growth factors within the past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
ASIA motor score | From enrollment to the end of treatment at 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fouad K, Popovich PG, Kopp MA, Schwab JM. The neuroanatomical-functional paradox in spinal cord injury. Nat Rev Neurol. 2021 Jan;17(1):53-62. doi: 10.1038/s41582-020-00436-x. Epub 2020 Dec 11. PMID 33311711
- [Result] Yang F, Zhang R, Xu J, Du J, Leng S, Zhang L, Huang D. Comparative Effects of Concentrated Growth Factors on the Biological Characteristics of Periodontal Ligament Cells and Stem Cells from Apical Papilla. J Endod. 2022 Aug;48(8):1029-1037. doi: 10.1016/j.joen.2022.05.001. Epub 2022 May 8. PMID 35545146
- [Result] Hu T, Zhang H, Yu W, Yu X, Li Z, He L. The Combination of Concentrated Growth Factor and Adipose-Derived Stem Cell Sheet Repairs Skull Defects in Rats. Tissue Eng Regen Med. 2021 Oct;18(5):905-913. doi: 10.1007/s13770-021-00371-y. Epub 2021 Jul 24. PMID 34302696
- [Result] Noh KC, Liu XN, Zhuan Z, Yang CJ, Kim YT, Lee GW, Choi KH, Kim KO. Leukocyte-Poor Platelet-Rich Plasma-Derived Growth Factors Enhance Human Fibroblast Proliferation In Vitro. Clin Orthop Surg. 2018 Jun;10(2):240-247. doi: 10.4055/cios.2018.10.2.240. Epub 2018 May 18. PMID 29854349
- [Result] Wang L, Wan M, Li Z, Zhong N, Liang D, Ge L. A comparative study of the effects of concentrated growth factors in two different forms on osteogenesis in vitro. Mol Med Rep. 2019 Aug;20(2):1039-1048. doi: 10.3892/mmr.2019.10313. Epub 2019 May 30. PMID 31173196
- [Result] Denapoli PM, Stilhano RS, Ingham SJ, Han SW, Abdalla RJ. Platelet-Rich Plasma in a Murine Model: Leukocytes, Growth Factors, Flt-1, and Muscle Healing. Am J Sports Med. 2016 Aug;44(8):1962-71. doi: 10.1177/0363546516646100. Epub 2016 May 23. PMID 27217525
- [Result] Christgau M, Moder D, Hiller KA, Dada A, Schmitz G, Schmalz G. Growth factors and cytokines in autologous platelet concentrate and their correlation to periodontal regeneration outcomes. J Clin Periodontol. 2006 Nov;33(11):837-45. doi: 10.1111/j.1600-051X.2006.00991.x. PMID 17018133
- [Result] Schar MO, Diaz-Romero J, Kohl S, Zumstein MA, Nesic D. Platelet-rich concentrates differentially release growth factors and induce cell migration in vitro. Clin Orthop Relat Res. 2015 May;473(5):1635-43. doi: 10.1007/s11999-015-4192-2. PMID 25690170
- [Result] Tabatabaei F, Aghamohammadi Z, Tayebi L. In vitro and in vivo effects of concentrated growth factor on cells and tissues. J Biomed Mater Res A. 2020 Jun;108(6):1338-1350. doi: 10.1002/jbm.a.36906. Epub 2020 Feb 28. PMID 32090458
- [Result] Courtine G, Sofroniew MV. Spinal cord repair: advances in biology and technology. Nat Med. 2019 Jun;25(6):898-908. doi: 10.1038/s41591-019-0475-6. Epub 2019 Jun 3. PMID 31160817
- [Result] Hutson TH, Di Giovanni S. The translational landscape in spinal cord injury: focus on neuroplasticity and regeneration. Nat Rev Neurol. 2019 Dec;15(12):732-745. doi: 10.1038/s41582-019-0280-3. Epub 2019 Nov 14. PMID 31728042
- [Result] Lu Y, Shang Z, Zhang W, Hu X, Shen R, Zhang K, Zhang Y, Zhang L, Liu B, Pang M, Rong L. Global, regional, and national burden of spinal cord injury from 1990 to 2021 and projections for 2050: A systematic analysis for the Global Burden of Disease 2021 study. Ageing Res Rev. 2025 Jan;103:102598. doi: 10.1016/j.arr.2024.102598. Epub 2024 Nov 26. PMID 39603465
- [Result] Pedro KM, Fehlings MG. Progress and future directions in spinal cord injury trials. Lancet Neurol. 2025 Jan;24(1):3-5. doi: 10.1016/S1474-4422(24)00482-4. No abstract available. PMID 39706629